CLINICAL TRIAL: NCT00252174
Title: Phase II Dose-response Pilot Study of 3,4-methylenedioxymethamphetamine (MDMA)-Assisted Psychotherapy in Subjects With Anxiety Associated With Advanced-stage Cancer.
Brief Title: MDMA-assisted Therapy in People With Anxiety Related to Advanced Stage Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funds and insufficient patient population for study enrollment.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Principal Investigator, John H. Halpern, MD, Director, Laboratory for Integrative Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 76,770
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Anxiety Disorder; Cancer
Keywords: MDMA; cancer; anxiety; psychotherapy; quality of life
MeSH Terms: conditions — Anxiety Disorders; Neoplasms | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Stage 1 Active methylenedioxymethamphetamine & psychotherapy (Experimental): 8 subjects will receive full or nearly full doses of MDMA in Stage 1 and do not continue to participate into Stage 2.
  Interventions: Drug: Stage 1 Active Methylenedioxymethamphetamine; Behavioral: Psychotherapy
- Stage 1 low dose methylenedioxymethamphetamine & Psychotherapy (Active Comparator): 4 individuals will receive sub-threshold to threshold minimal doses of MDMA in Stage I
  Interventions: Drug: Stage 1 Low dose Methylenedioxymethamphetamine; Behavioral: Psychotherapy
- Stage 2 Active methylenedioxymethamphetamine & Psychotherapy (Experimental): The 4 subjects assigned in Stage I to the control arm will have the option to continue into Stage 2 to repeat the experimental procedures of Stage I but with open-label MDMA at the near-full to full dosage strength.
  Interventions: Behavioral: Psychotherapy; Drug: Stage 2 Active Methylenedioxymethamphetamine

INTERVENTIONS:
Drug: Stage 1 Active Methylenedioxymethamphetamine — Dosage form: capsule
  Dosage frequency and duration for the treatment arm (8 subjects in Stage 1 and the other 4 subjects in Stage 1 who may continue into Stage 2):
  Session 1: 83.3mg followed 2.5 hours later with optional 41.7 mg for total of 125mg Session 2 (two to three weeks later): 125mg followed 2.5 hours later with optional 62.5mg for total of 187.5 mg.
  Arms: Stage 1 Active methylenedioxymethamphetamine & psychotherapy
Drug: Stage 1 Low dose Methylenedioxymethamphetamine — Drug:
  Dosage form: capsule
  Dosage frequency and duration for the control arm (4 subjects):
  Session 1: 25 mg followed 2.5 hours later with optional 12.5 mg for total of 37.5 g Session 2 (two to three weeks later): 25 mg followed 2.5 hours later with optional 12.5mg for total of 37.5mg.
  Arms: Stage 1 low dose methylenedioxymethamphetamine & Psychotherapy
Behavioral: Psychotherapy — Psychotherapy conducted with low or active dose MDMA
Drug: Stage 2 Active Methylenedioxymethamphetamine — Administered open label Dosage form: capsule
  Dosage frequency and duration for the treatment arm (8 subjects in Stage 1 and the other 4 subjects in Stage 1 who may continue into Stage 2):
  Session 1: 83.3mg followed 2.5 hours later with optional 41.7 mg for total of 125mg Session 2 (two to three weeks later): 125mg followed 2.5 hours later with optional 62.5mg for total of 187.5 mg.
  Arms: Stage 2 Active methylenedioxymethamphetamine & Psychotherapy

SUMMARY:
This is a pilot study intended to find out if 3,4-methylenedioxymethamphetamine (MDMA) is safe and can help people with advanced stage cancer and anxiety arising from the cancer diagnosis.

DETAILED DESCRIPTION:
People who learn they have cancer can feel frightened, upset and depressed, and a diagnosis of advanced stage cancer can generate intense anxiety. People with advanced stage cancer may be anxious about their deteriorating health and the nearness of death, disruption in their close relationships caused by current or future changes in health, and grief for the life planned and expected prior to learning they had advanced stage cancer. There are treatments for reducing intense anxiety, such as Valium and related drugs, but these drugs have unwanted side effects that may be especially distressing for people already taking medication for pain control and seeking to remain clear-headed.

3,4-methylenedioxymethamphetamine (MDMA) is a drug that can produce effects uniquely suited to reducing anxiety for people with anxiety arising from a cancer diagnosis. MDMA has been hypothesized to belong to a class of drugs, called entactogens, that produce feelings of closeness to others, empathy, wellbeing, and insightfulness. Currently, MDMA is scheduled (illegal) and cannot be used outside of research studies like this one. However, prior to its being made illegal, some psychotherapists treated people with cancer or other terminal illnesses with MDMA-assisted psychotherapy, and they reported a reduction in anxiety and improved quality of life.

This study will examine the effects of MDMA-assisted psychotherapy in 12 people aged 18 or older who have received a diagnosis of advanced stage cancer (usually meaning inoperable and with metastases) who have anxiety as a result of this diagnosis that is either not helped by conventional anti-anxiety medication (such as Xanax or Valium), or who do not wish to take these medications because of their side effects. In Stage 1, all study subjects will receive an initial dose of MDMA followed by a second (supplemental) dose approximately two and a half hours later if the initial dose does not produce any problems. Eight of twelve study subjects will get 83.3 mg MDMA followed by 47.1 mg the first time, and 125 mg followed by 67.5 mg the second time. Four of twelve study subjects will receive 25 mg followed by 12.5 mg MDMA. Whether a person receives low doses or full doses of MDMA will be decided at random, as if by coin toss, and none of the researchers will know which dose of MDMA a person will get in Stage 1. The four subjects who received the lower doses of MDMA in Stage 1 may continue to participate into Stage 2 in which they repeat the study except that they will receive open-label 83.3 mg MDMA followed by 47.1 mg the first time, and 125 mg followed by 67.5 mg the second time. The eight participants in Stage 1 who had MDMA-assisted psychotherapy sessions at these higher dose strengths will not continue into Stage 2. The Stage 2 study extension will provide potential additional data on the MDMA doses being evaluated without having to recruit additional subjects.

For Stage 1, the study will last 14 weeks (about three and a half months). All study participants will have six (6) hour-long psychotherapy sessions and two (2) MDMA-assisted psychotherapy sessions lasting six to eight hours and requiring an overnight stay at the treatment facilities. The ordinary and MDMA-assisted sessions will be conducted by the same therapists. For the four subjects continuing into Stage 2, the study will last an additional 10 weeks (about two and a half months) with additional six (6) hour-long psychotherapy sessions and two (2) MDMA-assisted psychotherapy sessions lasting six to eight hours and requiring an overnight stay at the treatment facilities.

People enrolled in the study can continue taking anti-anxiety medications, but cannot take any other psychiatric medications for the entire course of the study. They can take their usual pain control medications, but if they take more pain control medications than usual on the day of the MDMA-assisted session, they may have to delay or reschedule the session. People enrolled in this study will complete questionnaires about their anxiety and quality of life, and they will keep a daily diary where they write down how much anxiety and pain control medication they are using, and a daily record of the amount of pain they experience.

Anxiety and quality of life will be measured at the start of the study, before each sessions of MDMA-assisted therapy, one week after receiving MDMA-assisted therapy and once at the end of the study, 84 days after a person started the study (approximately two months after the second MDMA-assisted psychotherapy session; for Stages 1 and 2). All study subjects will also receive a second medical examination 36 days after the study has begun (and again 36 days after starting Stage 2). The medical examination will be performed at the Lahey Clinic Medical Center's Medical Oncology department or at McLean Hospital.

Study participants will not be paid for taking part in the study. We will pay for all tests and measures used to determine study eligibility. Transportation, if needed, will also be paid for by the study. MDMA-assisted sessions require overnight stay at McLean Hospital: we will provide overnight accommodations and all meals and snacks for the subject and a significant support person of the subject's choosing on those days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with advanced-stage cancer (usually meaning inoperable or incurable) with a life expectancy of less than 12 months.
* Anxiety as a result of cancer diagnosis
* Failure to respond adequately or at all to medication intended to reduce anxiety, or have refused to take anxiolytic medication.
* Completed or independently decided to end all direct cancer treatments, such as chemotherapy and radiation, two weeks prior to the first experimental (MDMA) session. If subjects wish to initiate or resume treatment for cancer at any point prior to the second experimental (MDMA) session, then they will be withdrawn from the study and will be asked to see the co-investigator oncologist for a final physical examination. Participants will not be withdrawn from the study if they initiate or resume treatment after the second experimental (MDMA) session. Those who are receiving cycles of cancer treatments for only palliative purposes (no longer for any curative reasons or to induce complete remission), may also be included in this study provided that they, as well, have completed their last cycle of treatment at least two weeks prior to the first experimental (MDMA) session and provided that they will not resume another cycle of treatment until after completion of the second experimental (MDMA) session. If a subject receiving palliative cancer treatment decides to receive a next cycle of this cancer treatment prior to the second experimental session, then, again, they will be withdrawn from the study. Participants will not be withdrawn from the study if they initiate or resume palliative cancer treatments after the second experimental (MDMA) session.
* Willing to commit to and follow all directions and restrictions relating to the study period
* Must be willing and able to discontinue use of psychiatric medication except that being used to treat anxiety. If still taking medication when enrolled to the study, medication will be discontinued long enough before the first MDMA-assisted psychotherapy session to avoid a drug-drug interaction
* Must be willing and able to stay overnight at the facility after each MDMA-assisted session.
* If seeing another psychotherapist, participants must be willing to give the principal investigator permission to communicate with him or her.
* Female participants of childbearing potential must have a negative pregnancy test and must agree to use an effective form of birth control.

Exclusion Criteria:

* People with a life expectancy of longer than 12 months
* Women who are pregnant or nursing, or of child bearing potential and are not practicing an effective means of birth control.
* People with any dissociative disorder, anorexia nervosa, bulimia nervosa, a primary psychotic disorder or affective disorder other than anxiety related to advanced stage cancer
* People diagnosed with abuse of or dependence on any substance (other than caffeine or nicotine) in the past 60 days.
* People with known primary or metastatic cancer of the CNS
* People with significant, unstable hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, that in the clinical judgment of the investigators poses too great a potential for side-effects.
* People with significant peripheral vascular disease, hepatic disease, renal insufficiency, or preexisting or past evidence of hyponatremia.
* People diagnosed with hypertension, even if well-controlled with medication. A systolic blood pressure of 140 or greater and/or a diastolic blood pressure of 90 or greater will exclude the potential participant from this study.
* People with liver enzyme values indicative of severely compromised hepatic (liver) function
* People who weigh less than 45 kg (98 lb)
* People reporting a history of use of "ecstasy" (illicit drug preparations purported to contain MDMA) at any time within the previous 3 months.
* People reasonably judged to present a serious suicide risk or who are likely to require psychiatric hospitalization during the course of the study
* People requiring psychotropic medication other than anxiolytic medication or for pain control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-02; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Halpern, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1, Active: 8 subjects will receive full or nearly full doses of MDMA in Stage 1 and do not continue to participate into Stage 2.
  3,4-methylenedioxymethamphetamine (MDMA): Dosage form: capsule
  Dosage frequency and duration for the treatment arm (8 subjects in Stage 1 and the other 4 subjects in Stage 1 who may continue into Stage 2):
  Session 1: 83.3mg followed 2.5 hours later with optional 41.7 mg for total of 125mg Session 2 (two to three weeks later): 125mg followed 2.5 hours later with optional 62.5mg for total of 187.5 mg.
- Stage 1, Control: 4 individuals will receive sub-threshold to threshold minimal doses of MDMA in Stage I
  3,4-methylenedioxymethamphetamine (MDMA): Drug: Dosage form: capsule
  Dosage frequency and duration for the control arm (4 subjects):
  Session 1: 25 mg followed 2.5 hours later with optional 12.5 mg for total of 37.5 g Session 2 (two to three weeks later): 25 mg followed 2.5 hours later with optional 12.5mg for total of 37.5mg.
- Stage 2, Active: The 4 subjects assigned in Stage I to the control arm will have the option to continue into Stage 2 to repeat the experimental procedures of Stage I but with open-label MDMA at the near-full to full dosage strength.
  3,4-methylenedioxymethamphetamine (MDMA): Dosage form: capsule
  Dosage frequency and duration for the treatment arm (8 subjects in Stage 1 and the other 4 subjects in Stage 1 who may continue into Stage 2):
  Session 1: 83.3mg followed 2.5 hours later with optional 41.7 mg for total of 125mg Session 2 (two to three weeks later): 125mg followed 2.5 hours later with optional 62.5mg for total of 187.5 mg.
Period: Overall Study
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Started | 0 (No subjects were randomized into Active Arm as only 2 subjects were randomized into the Control Arm.) | 2 (2 subjects entered the control arm in total) | 0 (No subjects entered Stage 2)
Completed | 0 | 1 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active | Total
Number analyzed (Participants) | 0 | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 |  | 0
  Between 18 and 65 years |  | 0 |  | 0
  >=65 years |  | 2 |  | 2
Age, Continuous [Mean (Full Range); unit: years] |  | 66 [65 to 67] |  | 66 [65 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 |  | 0
  Male |  | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  | 0
  Not Hispanic or Latino |  | 2 |  | 2
  Unknown or Not Reported |  | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0
  Asian |  | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0
  Black or African American |  | 0 |  | 0
  White |  | 2 |  | 2
  More than one race |  | 0 |  | 0
  Unknown or Not Reported |  | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Spielberger State-Trait Anxiety Inventory (STAI)
Description: Established self-report measure of anxiety containing a State and Trait subscale and scored on a four-point Likert scale. Scores for each subscale range from 10 to 40 and combined from 20 to 80 with higher scores indicative of greater anxiety.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Quality of Life - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Self-report instrument assessing quality of life with five functional scales, and nine symptom scales. Higher functional scores indicate better quality of life and higher symptom scores indicate poorer quality of life. Scales include "Yes" / "No" responses and four-point Likert scales, with transformations performed on scores so that all scale scores range from 0 to 100.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Anxiety - Hamilton Anxiety Rating Scale (HAM-A)
Description: standardized assessment of anxiety
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Quality of Life - Functional Assessment of Chronic Illness Therapy- Spiritual Well-being Scale (FACIT-Sp),Karnofsky Performance Rating Scale (KPRS), Memorial Symptom Assessment Scale (MSAS), Mini-Mental Status Exam (MMSE), Self-Expansiveness Level Form
Description: paper pencil tests capturing data on spiritual well-being, overall functioning living with cancer, psychiatric mental status, and on spiritual self-perception.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: Standardized interview assessing of depression, with higher scores indicative of greater depression. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Depression, Thoughts of Death - Schedule of Attitudes Toward Hastened Death (SAHD)
Description: standardized questions to evaluate extent of depression and thoughts of death.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Daily Use of Anxiolytics - Daily Diary
Description: daily log of anxiolytic medication usage.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Daily Experience of Pain - Visual Analog Pain Scale (VAPS)
Description: daily measure of self-reported pain.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: The Hospital Anxiety and Depression Scale (HADS)
Description: Standardized assessment of anxiety and depression consisting of a 7-item anxiety scale and a 7-item depression scale. Each scale score ranges from 0 to 21, with 0-7 being "normal" and 11-21 being "abnormal" [e.g. severely depressed or anxious]
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Daily Assessment of Anxiety - the Visual Analog Anxiety Scale (VAAS)
Description: Daily self-report measure for anxiety.
Time Frame: Obtained over the 3 months of active participation
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Beck Hopelessness Scale (BHI)
Description: Established self-report measure of depression and hopelessness, consisting of 20 true-false questions, with scores ranging from 0 to 20, with scores of 0-3 indicating minimal hopelessness and scores of 15-20 severe hopelessness.
Time Frame: Obtained over 3 months of study
Population: Data has been damaged/lost in a flood that destroyed the office that contained much of the primary source material
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Stage 1, Active | Stage 1, Control | Stage 2, Active
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes